CLINICAL TRIAL: NCT04726735
Title: Evaluation of PD-L1 Expression and Immune Infiltration in High-risk Non Muscle Invasive Bladder Cancer
Acronym: IMMUN VESSIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2018/55
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Bladder Cancer
Keywords: Non Muscle Invasive Bladder Cancer; Bacillus Calmette-Guerin; Programmed cell Death-Ligand protein 1; Programmed cell Death 1; Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — samples taken from 2007 to 2011 and stored in the tissue bank from Bordeaux hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with histologically documented normal bladder
  Interventions: Biological: Samples of bladder tissue
- Patients with histologically documented Non Muscle Invasive Bladder Cancer
  Interventions: Biological: Samples of bladder tissue
- Patients with histologically documented Muscle Invasive Bladder Cancer
  Interventions: Biological: Samples of bladder tissue

INTERVENTIONS:
Biological: Samples of bladder tissue — Samples of bladder tissue collected between 2007 and 2011.

SUMMARY:
Non-muscle-invasive bladder cancer (NMIBC) has a high rate of recurrence (60 to 70%) and progression (20 to 30%) to muscle-invasive bladder cancer (MIBC).

The local immunotherapy (intra-vesical Bacillus Calmette-Guerin (BCG) following transurethral resection of the bladder tumor (TURBT)) reduces significantly the risk of recurrence and progression as compared to observation or to intra-vesical chemotherapy.

Systemic immunotherapy with programmed death ligand-1 (PD-L1) or Programmed cell Death 1 (PD1) inhibitors has shown major efficacy in the treatment of patients with advanced/metastatic urothelial carcinoma who have progressed on platinum-based regimens of chemotherapy, or even in front line setting. In the field of NMIBC, immunotherapy using PD-L1 or PD1 inhibitors is under investigation but the frequency of PD-L1 expression has rarely been precisely described in the different subtypes.

The aim of this retrospective study is to investigate the expression of PD-L1 by different types of NMIBC.

The secondary objective is to characterize the immune contexture of NMIBC.

DETAILED DESCRIPTION:
Non-muscle-invasive bladder cancer (NMIBC) has a high rate of recurrence (60 to 70%) and progression (20 to 30%) to muscle-invasive bladder cancer (MIBC).

The local immunotherapy (intra-vesical Bacillus Calmette-Guerin (BCG) following transurethral resection of the bladder tumor (TURBT)) reduces significantly the risk of recurrence and progression as compared to observation or to intra-vesical chemotherapy.

Systemic immunotherapy with programmed death ligand-1 (PD-L1) or Programmed cell Death 1 (PD1) inhibitors has shown major efficacy in the treatment of patients with advanced/metastatic urothelial carcinoma who have progressed on platinum-based regimens of chemotherapy, or even in front line setting. In the field of NMIBC, immunotherapy using PD-L1 or PD1 inhibitors is under investigation but the frequency of PD-L1 expression has rarely been precisely described in the different subtypes.

The aim of this retrospective study is to investigate the expression of PD-L1 by different types of NMIBC.

The secondary objective is to characterize the immune contexture of NMIBC. The immunological contexture of NMIBC in comparison with normal bladder tissue and invasive bladder cancer will be deciphered. The objective is to determine immune signatures associated with response or relapse/progression, with and without immune treatments in NMIBC.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically documented normal bladder, NMIBC (Ta, T1, CIS) or MIBC stored in the tissue bank.

Samples collected from 2007 to 2011. 3 years follow-up is mandatory to assess the frequency of recurrences and progressions.

Exclusion Criteria:

* History of autoimmune disease
* Active tuberculosis
* Prior treatment with CD137 agonists, anti-programmed death-1 (PD-1), or anti-PD-L1 therapeutic antibody or pathway-targeting agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically documented normal bladder, NMIBC (Ta, T1, CIS) or MIBC stored in the tissue bank.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
PD-L1 status (positive or negative) of the tumor and tumor associated immune cells. | Day 1
  PD-L1 status will be considered positive if more than 25% of tumor cells exhibit membrane staining or immune cells present (ICP) >1% and immune cells (IC)+ >25% or ICP=1% and IC+ = 100%.
  PD-L1 status will be considered negative if none of the criteria for PD-L1 positive status are met.

SECONDARY OUTCOMES:
Descriptive analysis of the differential expression of all the following immune biomarkers in normal bladder tissue, NMIBC (Non Muscle Invasive Bladder Cancer) and MIBC (Muscle Invasive Bladder Cancer). | Day 1
  Descriptive statistics will be performed from clinical characteristics as mean values for categorical variables, or medians (range) for non-normal continuous variables.
Association of immune profile with recurrence and progression rates | Day 1
  Association between all variables will be analysed with t-test, Mann Whitney or ANOVA multiple comparison test. Correlation analysis will be performed with χ2 and Fischer exact test. Results will be considered significant if the p-value is <0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Talence, France

IPD SHARING:
Plan to Share IPD: No